CLINICAL TRIAL: NCT00591825
Title: An fMRI Study Investigating the Effects of Acute D-cycloserine Administration on Brain Activations and Cognitive Functioning in Spider Phobia.
Brief Title: fMRI Study Examining Effects of D-cycloserine in Specific Phobia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Collaborators: American Psychological Foundation (Other); American Psychological Association (Unknown)
Responsible Party: Principal Investigator, Cary Savage, Ph.D., Director, CHBN and John H. Wineinger Professor of Psychiatry and Behavioral Sciences, University of Kansas
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 10362; GCRC 0046 (Other: University of Kansas Medical Center); HSCL 15970 (Other: University of Kansas)
Record Dates: First submitted 2007-12-27; First posted 2008-01-11 (Estimated); Results first posted 2017-06-05 (Actual); Last update posted 2017-06-05 (Actual); Status verified 2017-06

CONDITIONS: Phobias
MeSH Terms: conditions — Phobic Disorders | interventions — Cycloserine; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Non-Phobic Control - Placebo (Placebo Comparator): Participants without phobia will be given one placebo administration.
  Interventions: Drug: Placebo
- Non-Phobic Control - DCS (Active Comparator): Participants without phobia will be given one D-cycloserine (DCS) administration of 100mg.
  Interventions: Drug: D-cycloserine
- Spider-phobic Placebo (Placebo Comparator): Participants with phobia will be given one placebo administration.
  Interventions: Drug: Placebo
- Spider-phobic DCS (Experimental): Participants with phobia will be given one D-cycloserine (DCS) administration of 100mg.
  Interventions: Drug: D-cycloserine

INTERVENTIONS:
Drug: D-cycloserine — D-cycloserine
  Other Names: Cycloserine
  Arms: Non-Phobic Control - DCS; Spider-phobic DCS
Drug: Placebo — Placebo
  Other Names: Sugar pill
  Arms: Non-Phobic Control - Placebo; Spider-phobic Placebo

SUMMARY:
The research team hopes to use brain imaging and mental testing to learn more about specific phobias and the treatment of phobia. When given directly prior to therapy sessions, D-cycloserine has been shown to enhance the effects of therapy. This study hopes to identify reasons why D-cycloserine has this effect by measuring brain activity.

DETAILED DESCRIPTION:
Exposure and Response Prevention (ERP) therapy has become the treatment of choice for specific phobias. ERP involves systematic and repeated exposure to a feared or anxiety-provoking stimulus, leading to habituation and extinction of the fear response. Animal models of fear extinction have shown that acute administration of D-cycloserine (DCS) prior to exposure to a feared stimulus enhances extinction of that fear. A recent study in human subjects with height phobia (a specific phobia) has also demonstrated that DCS facilitates the effects of ERP therapy. Current theories postulate that DCS facilitates fear extinction by enhancing the learning process and increasing consolidation of memories, but the neural mechanisms underlying this process are not understood. The proposed research aims to elucidate these mechanisms by using fMRI to measure brain activation during 1) symptom provocation and verbal learning two hours post-medication, and 2)repeated symptom provocation and verbal recognition one week post-medication. This research will also examine the effects of DCS on cognitive functioning using neuropsychological testing both two house and one week post-medication.

ELIGIBILITY:
Inclusion Criteria:

* Right-handed
* Adults between 18 and 55 years of age
* Subjects in the phobic group will additionally meet diagnostic (DSM-IV) criteria for spider phobia.
* Individuals of both genders and all races will be included

Exclusion Criteria:

* Women who are breastfeeding or pregnant
* Individuals with medical conditions unsuitable for MR scanning
* Individuals reporting a history of epilepsy or seizures
* Individuals reporting an allergy to cycloserine
* Individuals diagnosed with asthma or who report previous anaphylactic reaction to insect stings/bites, medication, food, or other material and/or event
* Individuals reporting present or past diagnosis of a developmental disorder, neurological disorder, or head injury *Individuals found to have Axis I psychopathology as defined by the DSM-IV (other than spider phobia)
* Individuals currently taking any psychotropic medication

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2006-03; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cary Savage, PhD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Hoglund Brain Imaging Center, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Non-Phobic Control - Placebo: Participants without phobia given one administration placebo.
- Non-Phobic Control - DCS: Participants without phobia given one administration of 100 mg D-cycloserine (DCS).
- Spider-phobic Placebo: Participants with phobia given one administration of placebo.
- Spider-phobic DCS: Participants with phobia given one administration of 100 mg D-cycloserine (DCS).
Period: Overall Study
Arm/Group | Non-Phobic Control - Placebo | Non-Phobic Control - DCS | Spider-phobic Placebo | Spider-phobic DCS
Started | 14 | 13 | 13 | 14
Completed | 14 | 13 | 13 | 14
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Non-Phobic Control - Placebo: Participants without phobia given one administration of placebo.
- Total: Total of all reporting groups
Arm/Group | Non-Phobic Control - Placebo | Non-Phobic Control - DCS | Spider-phobic Placebo | Spider-phobic DCS | Total
Number analyzed (Participants) | 14 | 13 | 13 | 14 | 54
Age, Continuous [Mean (Standard Deviation); unit: years] | 23.09 (3.70) | 26.75 (9.09) | 26.00 (8.06) | 24.73 (6.65) | 25.65 (7.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 9 | 7 | 13 | 39
  Male | 4 | 4 | 6 | 1 | 15

OUTCOME MEASURES:

1. Primary Outcome: fMRI Brain Activations During Symptom Provocation
Description: Regions of interest (ROIs) were specified based on previous research and included amygdala, insula, dorsal anterior cingulate cortex (ACC), dorsolateral PFC (dlPFC), and hippocampus. Multiple regression analyses were used to examine differences in response between experimental conditions (spider versus butterfly images). For significant clusters of activation within ROIs, the average max percent signal change is reported. For other regions, the average max percent signal change is reported within a sphere centered at coordinates identified via previous research.
Time Frame: 2 Weeks
Population: There were 54 enrolled in the study. 8 subjects were excluded from fMRI analyses: 1 for claustrophobia, 3 for scanner artifact, 1 because of motion >3mm; 3 of paradigm-consistent motion which could not be corrected for.
Measure: Mean (Standard Deviation); unit: percent signal change
Groups:
- DCS Phobic: Participants with phobia who were randomized to the DCS group were given one administration of 100 mg D-cycloserine (DCS).
- DCS Control: Participants without phobia who were randomized to the DCS group were given one administration of 100 mg D-cycloserine (DCS).
- Placebo Phobic: Participants with phobia who were randomized to the Placebo group were given one administration of placebo.
- Placebo Control: Participants without phobia who were randomized to the Placebo group were given one administration of placebo.
Arm/Group | DCS Phobic | DCS Control | Placebo Phobic | Placebo Control
Number analyzed (Participants) | 11 | 12 | 12 | 11
percent signal change
  Left Insula Spider | .200 (.182) | .157 (.373) | -.013 (.167) | .036 (.095)
  Left Insula Butterfly | .012 (.139) | .021 (.376) | .092 (.162) | .079 (.147)
  Right Insula Spider | .107 (.190) | .174 (.287) | -.004 (.087) | .020 (.250)
  Right Insula Butterfly | .017 (.144) | .109 (.221) | .133 (.139) | .017 (.211)
  mid dorsal ACC Spider | .242 (.135) | .402 (.459) | .073 (.171) | .071 (.180)
  mid dorsal ACC Butterfly | .022 (.114) | .053 (.166) | .085 (.123) | -.059 (.244)
  Left dlPFC Spider | .250 (.183) | .122 (.361) | .019 (.118) | .278 (.300)
  Left dlPFC Butterfly | .031 (.122) | .076 (.372) | .035 (.154) | .075 (.435)
  Right dlPFC Spider | .384 (.286) | .521 (.676) | .301 (.349) | .038 (.464)
  Right dlPFC Butterfly | .150 (.203) | .431 (.585) | .249 (.420) | .110 (.310)
  Left amygdala Spider | .322 (.182) | .202 (.308) | .534 (.272) | .427 (.244)
  Left amygdala Butterfly | .127 (.139) | .149 (.137) | .254 (.157) | .098 (.299)
  Right amygdala Spider | .241 (.157) | .155 (.347) | .183 (.336) | .133 (.230)
  Right amygdala Butterfly | .082 (.157) | .181 (.244) | .203 (.216) | -.017 (.273)
  Left hippocampus Spider | .101 (.222) | .196 (.217) | .185 (.184) | .131 (.206)
  Left hippocampus Butterfly | .010 (.180) | .065 (.112) | .204 (.170) | .086 (.158)
  Right hippocampus Spider | .113 (.315) | .310 (.224) | .075 (.193) | .361 (.347)
  Right hippocampus Butterfly | .017 (.103) | .219 (.203) | .155 (.118) | .329 (.283)

2. Secondary Outcome: Cognitive Functioning Measured Using the Wechsler Memory Scale III (Logical Memory and Faces Subtests)
Description: This scale measures the learning and memory of functioning adults. Logical Memory I and II and Faces I and II subtests were administered to participants. The tasks measure verbal and visual memory, respectively. Scoring is based on the number of story details or faces correctly recalled during immediate (Logical Memory I, Faces I) and 30 minute delayed (Logical Memory II, Faces II) conditions. Total score ranges from 0-75 on Logical Memory I, 0-50 on Logical Memory II, 0-48 on Faces I, and 0-48 on Faces II. For all subtests, higher scores indicate better memory performance.
Time Frame: 2 Weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Spider-phobic DCS: Participants without phobia given one administration of 100 mg D-cycloserine.
Arm/Group | Non-Phobic Control - Placebo | Non-Phobic Control - DCS | Spider-phobic Placebo | Spider-phobic DCS
Number analyzed (Participants) | 14 | 13 | 13 | 14
units on a scale
  Logical Memory 1 | 51.93 (8.91) | 49 (9.24) | 52.69 (10.30) | 52.93 (7.56)
  Logical Memory 2 | 34.36 (6.67) | 32.46 (7.03) | 34.85 (8.21) | 35.43 (5.20)
  Faces 1 | 40.43 (3.2) | 41.85 (2.73) | 41 (4.28) | 42.07 (3.83)
  Faces 2 | 41.93 (2.09) | 41.62 (2.99) | 41.62 (3.43) | 42.07 (3.97)

3. Secondary Outcome: Cognitive Functioning Measured Using the Rey-Osterrieth Complex Figure Test (RCFT)
Description: The RCFT assesses the a person's ability to use cues to retrieve information. The test measures visuospatial construction and memory. A person is asked to draw a figure. The figure is broken down into 18 elements. The score is based on their presence, completeness, and correct placement. Each element is scored from 0-2. The Copy, Immediate, and Delay results are scored on a 36 point scale. The higher the score, the better the person performed on the test with a 0 being the minimum and 36 being the maximum score. The organization score is scored according to whether the participant drew five cohesive units of the figure together, for a range of 0-6 and a higher score indicating better organizational performance.
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Non-Phobic Control - Placebo | Non-Phobic Control - DCS | Spider-phobic Placebo | Spider-phobic DCS
Number analyzed (Participants) | 14 | 13 | 13 | 14
units on a scale
  Organization | 4.93 (1.33) | 4.92 (1.55) | 3.69 (1.97) | 4.14 (1.96)
  Copy | 34.68 (2.49) | 34.46 (3.53) | 34.46 (2.15) | 34.50 (1.95)
  Immediate | 26.54 (3.97) | 24.77 (6.66) | 26.17 (3.76) | 26.14 (5.46)
  Delay | 26.08 (3.81) | 23.35 (7.11) | 26.13 (2.57) | 25.64 (5.36)

4. Secondary Outcome: Cognitive Functioning Measured Using the Iowa Gambling Test
Description: This test measures a person's emotional decision making. Participants are presented with virtual decks of cards on a computer. Participants are told that each card they draw will "win" them game money. However, sometimes cards result in "losing" game money. The task includes 100 trials and the total score represents the number of cards drawn from "bad" decks as compared to "good" or safe decks. Thus, the score ranges from -100 to +100, with higher sores representing better performance.
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Non-Phobic Control - Placebo: Participants without phobia were given one administration placebo.
- Non-Phobic Control - DCS: Participants without phobia were given one administration 100 mg D-cycloserine (DCS).
- Spider-phobic Placebo: Participants with phobia were given one administration placebo.
- Spider-phobic DCS: Participants with phobia were given one administration 100 mg placebo.
Arm/Group | Non-Phobic Control - Placebo | Non-Phobic Control - DCS | Spider-phobic Placebo | Spider-phobic DCS
Number analyzed (Participants) | 14 | 13 | 13 | 14
units on a scale | 44.29 (23.68) | 32.62 (26.76) | 28.58 (21.89) | 21.85 (28.42)

5. Secondary Outcome: Cognitive Functioning Measured Using the Wisconsin Card Sorting Task
Description: The Wisconsin Card Sorting Task measures executive functioning and cognitive flexibility. The task uses a deck of 64 cards that the participant must sort according to specified rules. The test is stopped when when six sequences of 10 correct responses have been achieved, or after the deck has been completed twice, which provides a cumulative total of 128 trials. We report the number of errors on the task, which has a range of 0 -128, with a higher score representing worse performance.
Time Frame: 2 weeks
Population: Two subjects did not complete the test because they had previous exposure to the test.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Spider-phobic DCS: Participants with phobia were given one administration 100 mg D-cycloserine (DCS).
Arm/Group | Non-Phobic Control - Placebo | Non-Phobic Control - DCS | Spider-phobic Placebo | Spider-phobic DCS
Number analyzed (Participants) | 14 | 13 | 13 | 12
units on a scale | 13.29 (6.98) | 13.62 (7.65) | 18.23 (16.58) | 15.67 (9.33)

ADVERSE EVENTS:
Time Frame: At the end of each session, approximately 4-6 hours after drug administration. Participants were monitored through study completion, an average of 1 week.
Arm/Group | Non-Phobic Control - Placebo | Non-Phobic Control - DCS | Spider-phobic Placebo | Spider-phobic DCS
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/13 | 0/13 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/13 | 0/13 | 0/14
Other Adverse Events (participants affected / at risk) | 0/14 | 0/13 | 0/13 | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes